CLINICAL TRIAL: NCT02806466
Title: Risk Factors for Early Remodelling in Severe Asthma in Children
Acronym: P'tit-ASTHME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2010/20
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthmatic children (Active Comparator)
  Interventions: Procedure: Fiberoptic bronchoscopy
- Non-asthmatic children (Sham Comparator)
  Interventions: Procedure: Fiberoptic bronchoscopy

INTERVENTIONS:
Procedure: Fiberoptic bronchoscopy

SUMMARY:
* Background: Asthma is a frequent disease characterized by bronchial hyperresponsiveness, inflammation and remodeling. Consistent epidemiological data indicate that outcome of asthma in adults may be determined in early childhood. This may be due to bronchial remodeling, an abnormal repair process that contributes to the development of poorly reversible airway narrowing. It appears very early in the natural history of the disease and involves increased mass of bronchial smooth muscle (BSM). The mechanism of such an increase has been related with an increase in smooth muscle cell proliferation. Recently, we have demonstrated that in severe asthma, BSM increased proliferation is induced by an enhanced mitochondrial biogenesis. Moreover, we have also shown that immature human, non-asthmatic airway smooth muscle cells (ASMC) proliferate to a greater extent than normal adult ASMC, in a similar fashion to adult asthmatic ASMC. Immature ASMC may thus have great potential to stimulate airway remodeling. We thus hypothesized that remodeling is an early process and certain characteristics of ASMC in severe preschool asthma may predispose such children to persistent remodeling with airway obstruction later in life.
* Purpose: To investigate prognostic factors of airway remodeling in preschool children, with special attention to ASMC proliferation (mitochondrial mass & biogenesis).
* Methods: In the initial phase of the project, 75 severe asthmatic preschool children (<5 yr) will be prospectively recruited from the "CHU de Bordeaux" and the "CHU de Toulouse" according to the "Haute Autorité de Santé" criteria. Inclusion visit will include written informed consent, asthma control evaluation, clinical examination, lung function testing (exhaled NO, plethysmography), prick tests, chest X Ray and blood sample for total IgE levels. Bronchial specimens from all subjects will be obtained by fiberoptic bronchoscopy at visit 2. Airway remodeling will be evaluated by morphological analysis. After smooth muscle mitochondria will be analyzed by electronic microscopy & immunoblotting. Comparison between the 2 groups will be performed by unpaired t tests for parametric data and x2-tests for non-parametric data. In the second phase of the project, patients will then be followed-up till the age of 7-10 yrs, when another bronchoscopy with biopsies will be performed.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic children

* Parents (and possibly the child) who gave written informed consent.
* Affiliated with a social security scheme.
* Age from 1 to less than 5 years.
* Severe persistent asthma according to the criteria of the National Health Authority (Annex I) or NEW PROPOSED CRITERIA (adapted ATS (42)):

Major criteria (> 1) Asthma control in mild to moderate level requiring

1. A continuous or semi continuous (≥ 50% of the year) by oral corticosteroids
2. A treatment with high doses of inhaled corticosteroids (> 500 micrograms / day of Beclomethasone, or equivalent (> 400 micrograms / day of Budesonide,> 200 micrograms / day of Fluticasone) for at least 6 weeks.

And

minor criteria (> 2)

1. The need for an additional daily treatment (β2-agonists, long-acting, theophylline, anti-leukotrienes)
2. Symptoms that require taking daily or almost daily of β2-agonists of short action
3. persistent obstruction (FEV <80% PEF variability> 20%) (If reliable spirometry, usually> 5 years of age)
4. One or more seeking care in emergency / year
5. At least three short courses of oral corticosteroids / year
6. Rapid Increases caused by the decrease of 25% of the dose of oral corticosteroids or inhaled
7. ATCD of severe acute asthma who put in life-threatening

Non-asthmatic children

* Non asthmatic child with indication of endoscopy:

  * Any endoscopy for a disease without acute or chronic inflammation in the biopsy area (≥1 to <5 years (1st part): congenital stridor, double aortic arch, foreign body removal inhaled, ...; ≥ 7 to ≤ 10 years ( 2nd component): inhaled foreign body removal, ...).
  * Parents (and possibly the child) who gave written informed consent.
  * Affiliated with a social security scheme.
* Children not asthmatic postmortem (retrospective and prospective)

  * Age from 1 to under 5 (1st part) or aged 7 to 10 years (2nd part) on the death
  * Died without pulmonary pathology in the sampled area
* Non asthmatic child with thoracic surgery:

  * Age from 1 to under 5 (1st part) or aged 7 to 10 years (2nd part).
  * Subject with pulmonary pathology, requiring thoracic surgery lobectomy, non-inflammatory in the sampled area.
  * Parents (and possibly the child) who gave written informed consent.
  * Affiliated with a social security scheme.

Exclusion Criteria:

Asthmatic children:

* Subject having a severe exacerbation of asthmatic disease requiring hospitalization in the 3 weeks preceding their inclusion.
* exclusion period on topic compared to another protocol.
* Subject with significant co-morbidity associated with asthma not of any nature whatsoever
* bronchial malformations (exclusion criterion ex post).
* Subject with a dental infection, or nasopharyngeal airway (viral or bacterial) with fever (> 39 ° C) in the 4 weeks preceding the survey.
* chronic viral infections (hepatitis, HIV).
* non-specific inclusion criteria to endoscopy:
* Review of hemostasis abnormal,
* Subject with a heart condition,
* Subject is not fasted for over 6 hours.

Children without asthma:

* Non-asthmatic children with indication of endoscopy:

  * asthma diagnosed by a doctor.
  * exclusion period on topic compared to another protocol.
  * Subject with significant co-morbidity associated with asthma not of any nature whatsoever.
  * bronchial malformations (exclusion criterion ex post).
  * Subject with a dental infection, or nasopharyngeal airway (viral or bacterial) with fever (> 39 ° C) in the 4 weeks preceding the survey.
  * chronic viral infections (hepatitis, HIV).
  * non-specific inclusion criteria to endoscopy:
  * Review of hemostasis abnormal,
  * Subject with a heart condition,
  * Subject is not fasted for over 6 hours.
* Children postmortem non-asthmatics:

  * asthma diagnosed by a doctor.
  * Subject with a dental infection, or nasopharyngeal airway (viral or bacterial) with fever (> 39 ° C) within 4 weeks before sampling of tissue.
  * chronic viral infections (hepatitis, HIV).
* Non-asthmatic children with thoracic surgery:

  * asthma diagnosed by a doctor.
  * exclusion period on topic compared to another protocol.
  * Subject with a dental infection, or nasopharyngeal airway (viral or bacterial) with fever (> 39 ° C) within 4 weeks before sampling of tissue.
  * chronic viral infections (hepatitis, HIV).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Airway remodeling (distance from the reticular membrane to the smooth muscle). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: MICHAEL FAYON, Professor, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux, Aquitaine
  - Hôpital des Enfants, Toulouse, Occitanie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayon M, Beaufils F, Esteves P, Campagnac M, Maurat E, Michelet M, Siao-Him-Fa V, Lavrand F, Simon G, Begueret H, Berger P; P'tit Asthme Study Group. Bronchial Remodeling-based Latent Class Analysis Predicts Exacerbations in Severe Preschool Wheezers. Am J Respir Crit Care Med. 2023 Feb 15;207(4):416-426. doi: 10.1164/rccm.202205-0913OC. PMID 36108144